CLINICAL TRIAL: NCT06664567
Title: Impact of a Proactive Strategy of General Practitioners on CRC Screening: a Registry-based Cluster-based Randomized Controlled Trial
Brief Title: Impact of a Proactive Strategy of General Practitioners on CRC Screening
Acronym: DECORE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2021/64
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer screening; general practitioner; social health inequalities
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Systematic provision of screening tests by GPs: The general practitioner systematically delivers the screening kit with justification and modalities of realization at an even age between 50 and 74 years to the patient who comes to consult for whatever reason, who is at intermediate risk of colorectal cancer and who falls under the generalized screening. The practitioner is helped in his approach by an initial training in the identification of the age, delivery of a poster, a study sheet, stickers and goodies, sending a quarterly letter on the progress of the study and contact with the coordination team.
  Interventions: Behavioral: Colorectal cancer screening test
- Delivery of screening test according to GP's usual practice: the GP will issue the CRC screening kit in accordance with his/her usual practice.
  Interventions: Behavioral: Colorectal cancer screening test

INTERVENTIONS:
Behavioral: Colorectal cancer screening test — delivery of colorectal cancer screening test by GP

SUMMARY:
In this registry-based cluster randomized controlled trial, we will assess the impact of a proactive strategy of general practitioners (GP) who will systematically provide screening kits of colorectal cancer (CRC) to all patients of even age (50, 52, 54...up to 74 years) versus usual practice where the eligible population receive an invitation letter to visit the general practitioner and receive the screening kit.

DETAILED DESCRIPTION:
Colorectal cancer is one of the leading causes of cancer and death in France in both men and women. The generalized screening rate is about 30% in France, far from the expected 65%, despite the fact that screening is free and a letter of invitation is sent to the individual's home, and despite the financial incentives provided to the practitioner. Different studies have looked for the causes of non-implementation by the individual: negligence, "dirty"; forgetfulness, and the practitioner: organizational problem, communication problem. A few intervention studies have been carried out with little success: sending the invitation to the individual's home, sending a letter of reminder, sending a letter of general information on screening to the practitioner, sending the list of patients who have not taken the test to the practitioner allows for a few percent improvement in screening. In this registry-based cluster randomized controlled trial, we will assess the impact of a proactive strategy of general practitioners who will systematically provide screening kits of colorectal cancer to all patients of even age (50, 52, 54 years...up to 74 years) versus usual practice where the eligible population receive an invitation letter to visit the general practitioner and receive the screening kit. The screening rate will be calculated for each arm at the end of the 2-year study with data from the health insurance.

ELIGIBILITY:
inclusion criteria:

- medical practices in Aquitaine region and their visiting patients eligible for colorectal cancer screening individuals aged between 50 and 74 years at intermediate risk of colorectal cancer).

Exclusion criteria:

* medical practices with less than five individual eligible for colorectal cancer screening.
* visiting patients aged less than 50 years or more than 74 years or at high or very high risk of colorectal cancer.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient between 50 and 74 years old
Sampling Method: Probability Sample
Enrollment: 26260 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Participation rate in CRC screening | 2 years after the start of protocol
  The primary endpoint of this trial is the rate of participation rate in CRC screening in the eligible patient population grouped with or without intervention. This criterion will be measured by retrospective analysis of retrospective analysis of National Health Data System data.

SECONDARY OUTCOMES:
Positive test results | 2 years after the start of protocol
  Rate of patients with positive test results
Positive test at an early stage | 2 years after the start of protocol
  rate of patients tested positive at an early stage
Positive test at a last stage | 2 years after the start of protocol
  rate of patients testing positive at a late stage